CLINICAL TRIAL: NCT03661489
Title: Phase III Confirmatory Efficacy and Safety Trial of Remimazolam (CNS7056) Compared With Propofol for Intravenous Anesthesia During Elective Surgery in ASA Class III/IV Patients
Brief Title: Efficacy and Safety of Remimazolam (CNS7056) Compared to Propofol for Intravenous Anesthesia During Elective Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Paion UK Ltd. (Industry)
Collaborators: ORION Clinical Services (Industry); Simbec Research (Industry); Creative Clinical Research GmbH (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CNS7056-022
Record Dates: First submitted 2018-09-03; First posted 2018-09-07 (Actual); Last update posted 2020-05-28 (Actual); Status verified 2020-05

CONDITIONS: Anesthesia, Intravenous
Keywords: remimazolam
MeSH Terms: interventions — remimazolam; Propofol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intravenous Remimazolam 50 mg (Experimental): For induction of general anesthesia, remimazolam is co-administered with remifentanil for analgesia and with a muscle relaxant as necessary.
  For maintenance of general anesthesia remimazolam is titrated to effect. Administration of boluses of remimazolam is allowed. Remifentanil is continued and/or titrated. Boluses of muscle relaxants are given throughout the surgical procedure as needed.
  Interventions: Drug: Remimazolam
- Intravenous Propofol 2% (Active Comparator): For induction of general anesthesia, propofol is co-administered with remifentanil for analgesia and with a muscle relaxant as necessary.
  For maintenance of general anesthesia propofol is titrated to effect. Administration of boluses of propofol is allowed. Remifentanil is continued and/or titrated. Boluses of muscle relaxants are given throughout the surgical procedure as needed.
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Remimazolam — For induction and maintenance of general anesthesia
  Arms: Intravenous Remimazolam 50 mg
Drug: Propofol — For induction and maintenance of general anesthesia
  Arms: Intravenous Propofol 2%

SUMMARY:
A phase III confirmatory trial evaluating the efficacy and safety of remimazolam (CNS7056) compared to propofol for intravenous anesthesia during elective surgery in ASA Class III/IV patients.

DETAILED DESCRIPTION:
This is a Phase III single-blind, randomized, controlled, non-inferiority multi-center trial in American Society of Anesthesiologists (ASA) Class III/IV patients undergoing elective surgery, comparing remimazolam to propofol for induction and maintenance of intravenous anesthesia. In accordance with general anesthetic standard regimen, remimazolam or propofol, will be administered together with remifentanil as analgesic agent, and with a neuromuscular blocker to facilitate intubation and achieve muscle relaxation

ELIGIBILITY:
Inclusion criteria

* Male or female ASA III/IV patients at least 18 years old, scheduled for an elective surgical procedure of a minimum duration of approximately 90 minutes under general anesthesia (GA) and planned to be extubated immediately post-operatively.
* Total intravenous GA with the requirement for mechanical ventilation via endotracheal tube and necessary invasive blood pressure (BP) monitoring either due to severity of illness, severity of concomitant diseases, type of surgery or decisions of the anesthesia staff.
* Patients scheduled to stay in the hospital long enough after the surgical procedure to perform all trial follow-up procedures (~1 day)
* For female patients of childbearing potential: Negative result of a pregnancy test taken shortly before the start of the administration of the IMP as well as consent to use highly effective birth control from the last menstrual cycle prior to the start of the IMP until the end of the trial follow-up procedures. Highly effective methods of birth control include:

  * Combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation: oral, intravaginal and transdermal
  * Progestogen-only hormonal contraception associated with inhibition of ovulation: oral, injectable and implantable
  * Intrauterine device (IUD)
  * Intrauterine hormone-releasing system (IUS)
  * Bilateral tubal occlusion
  * Vasectomised partner (provided that the partner is the sole sexual partner of the female patient of childbearing potential and that the vasectomised partner has received medical assessment of the surgical success)
  * Sexual abstinence (this method is not acceptable in Switzerland)

Women who had their last menstruation at least two years ago or who underwent surgical interventions (surgical birth control, bilateral oophorectomy, hysterectomy, etc.) are regarded as having no childbearing potential

Exclusion criteria

* Patients scheduled for spinal anesthesia, epidural anesthesia (central neuraxial anesthesia) or regional anesthesia. The placement of a peridural catheter with a test dose application of a local anesthetic drug (up to 5 mL) to verify correct positioning to achieve post-operative analgesia and the regional administration of local anesthetic for post-operative analgesia after wound closure is accepted.
* Patients undergoing transplant surgery, cardiac surgery, or intracranial neurosurgery, patients which have to be in prone position for surgery, emergency surgery, or any surgical procedure with the need for or scheduled for post-operative ventilator support.
* Patients undergoing surgical procedures that require keeping the BP at a high level, e.g. surgical procedures in beach chair position
* Patients with severe hypertension, i.e., one baseline result of systolic BP 200 mmHg or more and / or diastolic BP of 120 mmHg or more. Baseline is defined as the time after signature of the informed consent form (ICF) and before arrival in the operating room (OR) suite.
* Patients with total bilirubin of ≥3.0 mg/dL or ≥3 times increase in aspartate aminotransferase (ASAT) or alanine aminotransferase (ALAT) than the institutional reference range in laboratory tests, or any other laboratory results that make the patient unsuitable for the trial. All laboratory tests relevant for subject's enrolment must be performed within 7 days prior to start of IMP*

  * If the screening samples for the central laboratory were taken earlier than within the last 7 days prior to start of IMP, the lab parameters relevant for subject's enrolment are to be determined in a local laboratory within 7 days prior to start of IMP. If results from samples taken within 7 days prior to the start of the IMP/the surgery from a local laboratory are available, these can be used. If no results from the last 7 days prior to the start of the IMP/the surgery are available, samples need to be taken for the purpose of this trial and to be analysed in a local laboratory.
* Patients with end stage renal disease (ESRD) requiring scheduled dialysis
* Patients with known anaphylactic reactions to benzodiazepines, propofol, opioid analgesics, non-steroidal anti-inflammatory drugs (NSAIDs), dextran, neuromuscular blocking agents, flumazenil, naloxone, or other anesthetic agents, or a medical condition such that these agents are contraindicated (according to local label)
* Presence of acute alcoholic or illicit drug intoxication, shock or coma state
* Known current dependency from central nervous system depressant drugs or alcohol
* Patients with gastroparesis or delayed gastric emptying, gastric reflux or any other increased risk for gastric aspiration
* Patients with an anticipated (small mouth opening, impaired neck movement, goitre, head and neck tumours or any other anatomical reason) or known airway difficulties or with known difficulties in airway maintenance or mask ventilation
* Patients in whom Narcotrend (NCT) may not provide reliable results due to organic defect of the brain or forehead, or any neurologic disease interfering with the EEG monitoring
* Patients on treatment with valproate
* Any pregnant or breast-feeding patient
* Patients who participated in any clinical trial within 30 days or 5 times the half-life of the drug under investigation, whichever is longer, prior to the beginning of administration of the IMP. Exception: Non-interventional trials as defined in the European Clinical Trials Directive 2001/20/EC: A trial where the medicinal product(s) is (are) prescribed in the usual manner in accordance with the terms of the marketing authorisation. The assignment of the patient to a particular therapeutic strategy is not decided in advance by a trial protocol but falls within current practice and the prescription of the medicine is clearly separated from the decision to include the patient in the study. No additional diagnostic or monitoring procedures shall be applied to the patients and epidemiological methods should be used for the analysis of the collected data.
* Any patient judged to lack the ability to give informed consent or perform the trial assessments (e.g., due to dementia)
* Any patient judged by the Principal Investigator (PI) or Sub-Investigator to be inappropriate for the subject for any other reason

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 469 (Actual)
Dates: Start 2018-07-24 (Actual); Primary Completion 2020-04-02 (Actual); Study Completion 2020-04-02 (Actual)

PRIMARY OUTCOMES:
Percentage (%) of time of Narcotrend Index (NCI) values ≤ 60 during maintenance phase of general anesthesia (defined as time between the first skin incision and the completion of the last skin suture) | maintenance phase of general anesthesia (time between the first skin incision and the completion of the last skin suture)
  The primary efficacy endpoint (PEP) is the anesthetic effect of remimazolam and propofol assessed as percent (%) of time of NCI ≤60 during the maintenance phase of general anesthesia

SECONDARY OUTCOMES:
Number of events of critical decrease(s) in mean arterial blood pressure (MAP) | From start of Investigational Medicinal Product (IMP) administration until 15 minutes after first skin incision
  For this endpoint, each event from the following categories will be counted and summed up per patient:
  * Incidence of MAP dropping below 65 mmHg for at least 1 minute duration
  * Incidence of a MAP decrease of more than 20% below the calculated (mean) baseline MAP value for at least 1 minute duration
  * Incidence of a MAP decrease of more than 30% below the calculated (mean) baseline MAP value for at least 1 minute duration
  * Number of norepinephrine boluses (0.01 mg) required or, if an infusion is used to maintain MAP equal to or above 65 mmHg, then each time interval of 2 minutes duration of continuous norepinephrine infusion will be counted as one event.

OTHER OUTCOMES:
Percentage of time of NCI ≤60 and ≥40 during the maintenance phase | During the maintenance phase of general anesthesia: from first skin incision to last skin suture
  Adherence to a pre-defined corridor to avoid sedation being too light or being too deep
Time from start of IMP administration to loss of consciousness | During induction of general anesthesia
  Loss of consciousness is defined as modified observer's assessment of alertness / sedation = 0
Time from stop of IMP to end of extubation | During recovery phase of general anesthesia
  Extubation is defined as the precise time (hh:mm) by when the tracheal tube used for the mechanical ventilation is removed
Time from stop of IMP to Modified Aldrete Score = 10 | During recovery phase of general anesthesia
  The time by when full recovery is reached defined as the time by when the Modified Aldrete Score is 10 for the first time
Delirium assessed by the Nursing Delirium Screening Scale (Nu-DESC) | During Screening, shortly before starting IMP (in the preparation period), in the Recovery Period and during Follow-up (up to 1 week after the end of the surgery)
  Any appearance of symptoms indicating delirium will be captured using the Nu-DESC

CONTACTS AND LOCATIONS:
Overall Officials: Jörg Fechner, Prof. Dr., Principal Investigator — University Erlangen-Nürnberg
Locations (1):
- University of Erlangen, Erlangen, Bavaria, Germany

REFERENCES:
- [Background] Antonik LJ, Goldwater DR, Kilpatrick GJ, Tilbrook GS, Borkett KM. A placebo- and midazolam-controlled phase I single ascending-dose study evaluating the safety, pharmacokinetics, and pharmacodynamics of remimazolam (CNS 7056): Part I. Safety, efficacy, and basic pharmacokinetics. Anesth Analg. 2012 Aug;115(2):274-83. doi: 10.1213/ANE.0b013e31823f0c28. Epub 2011 Dec 20. PMID 22190555
- [Background] Wiltshire HR, Kilpatrick GJ, Tilbrook GS, Borkett KM. A placebo- and midazolam-controlled phase I single ascending-dose study evaluating the safety, pharmacokinetics, and pharmacodynamics of remimazolam (CNS 7056): Part II. Population pharmacokinetic and pharmacodynamic modeling and simulation. Anesth Analg. 2012 Aug;115(2):284-96. doi: 10.1213/ANE.0b013e318241f68a. Epub 2012 Jan 16. PMID 22253270